CLINICAL TRIAL: NCT05661448
Title: Promoting Cognitive Health in Schizophrenia: A National Collaborative Effort to Implement Online Psychological Interventions
Brief Title: Promoting Cognitive Health in Schizophrenia
Acronym: iCogCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McGill University (Other)
Responsible Party: Principal Investigator, Martin Lepage, James McGill Professor, Douglas Mental Health University Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iCogCA
Record Dates: First submitted 2022-11-01; First posted 2022-12-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Cognition
Keywords: intervention; cognitive remediation; metacognition; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: A non-randomized concurrent control design (NRCC) is proposed and will allow for a comparison between the two interventions using one (e.g., CR) as the active control for the other (e.g., MCT) and vice-versa, on intervention-specific primary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive remediation (Experimental): CR was developed by Dr. Bowie (PI). Approximately 60% of CR sessions are spent on cognitive training activities, 20% on developing, monitoring, and flexibly adjusting problem-solving strategies, and 20% on transfer activities. Transfer includes discussing and role-playing how cognitive skills and strategies are applied in everyday life and teaches potential compensatory strategies for overcoming cognitive challenges. Targeted cognitive domains are processing speed, attention, memory, and executive functions, which are all commonly impaired in psychosis. The manual includes 1.5-hour sessions and uses Brain Training Pro and will be offered over an 8-week period. Zoom Health will be used for group transfer activities.
  Interventions: Behavioral: Cognitive remediation
- MetaCognitive Training (Experimental): MCT, developed by Drs. Moritz (co-applicant) and Woodward (PI), is based in the theoretical foundations of CBT, but targets the biases underlying symptoms rather than symptoms directly. MCT includes eight modules targeting common cognitive errors and reasoning biases in schizophrenia that have, through decades of research, been shown to contribute to delusions (e.g., jumping to conclusions). MCT will be offered to groups of up to 8 participants over 12 sessions of 45-60 min each (two per week) through Zoom Health. Session aims include raising participants' awareness of distortions and prompting them to critically reflect on, expand upon, and change their current repertoire of problem-solving strategies.
  Interventions: Behavioral: MetaCognitive Training

INTERVENTIONS:
Behavioral: Cognitive remediation — The goal of this program is to improve performance on cognitive domains known to hinder functioning. It aims to promote positive attitudes towards learning and facilitate the development of independent learning skills to foster competence and confidence. Another aim is to increase patients' awareness of their cognitive strengths and weaknesses and their own problem solving strategies.
  Other Names: Action-Based Cognitive Remediation
  Arms: Cognitive remediation
Behavioral: MetaCognitive Training — The metacognitive training (MCT) program is based on the theoretical foundations of cognitive models of schizophrenia but employs a slightly different focus in its therapeutic approach targeting the specific cognitive biases underlying delusions. The modules aim to raise awareness of these biases and prompts participants to critically reflect on and update their problem-solving repertoire.
  Arms: MetaCognitive Training

SUMMARY:
The goal of this clinical trial is to effectively implement virtually-delivered interventions in mental health institutions nationwide to improve the cognitive health of individuals living with schizophrenia. The main objectives are:

* To determine the clinical effectiveness of two virtual cognitive health interventions (i.e., Action-Based Cognitive Remediation or MetaCognitive Training).
* To evaluate our implementation strategy involving the virtual delivery of cognitive health interventions combined with a digital learning platform to train mental health practitioners.

Participants will be assessed for the severity of symptoms, cognitive performance, and overall functioning before and after receiving the intervention. Qualitative interviews will also be conducted with participants and therapists to evaluate the implementation strategies.

DETAILED DESCRIPTION:
In Canada, few individuals with psychotic disorders have access to online psychosocial therapies integrated with the care they receive from the public mental health care system. There is thus an urgent need for pragmatic trials, conducted in diversified settings, on the effectiveness and implementation of technology- enabled psychosocial interventions in this population. Even at the respective sites of the investigators, such interventions are predominately offered within the context of research and not as a clinical service. The investigators propose a hybrid effectiveness-implementation trial relying on digital technology to facilitate the rapid adoption of high- quality psychosocial interventions in five distinct care settings (Douglas Institute, Royal Institute of Mental Health Research, Kingston Health Science Centre, Ontario Shores Centre for Mental Health Sciences and Vancouver Coastal Health/UBC). Each site provides a unique environment to promote the uptake of interventions; all have a track-record of integrated clinical infrastructure for psychological interventions and access to large cohorts of potential participants (n>6000). These sites have all been providing psychological interventions for schizophrenia for several years and have the necessary infrastructure to provide virtual care.

Considering that both proposed cognitive health interventions are well established, the investigators are proposing a hybrid effectiveness-implementation design, Type 2 which is ideal when studying interventions that already have evidence of effectiveness in other settings or populations and that seek to determine feasibility and utility of an implementation strategy. Such designs are now commonly used to move evidence-based behavioral interventions into real care environments as they address the need to confirm clinical effectiveness while targeting the methods and procedures necessary to deliver and sustain such interventions in real-world care settings.

Objective 1: To determine the clinical effectiveness of two virtual cognitive health interventions. The investigators will use a non-randomized concurrent control design (NRCC) in which one intervention (e.g., CR) acts as the active control for the other (e.g., MCT) and vice-versa, on intervention-specific primary outcomes. The investigators hypothesize that participation in CR will specifically improve cognitive capacity (i.e., increase performance on measures of memory, executive functions, attention, etc.) whereas participation in MCT will specifically improve cognitive biases, per the objective standard measures described below. Moreover, participation in either intervention will be associated with improvement in symptomatology, reduced social isolation and greater functioning at post-intervention and maintained at 1 month follow-up. The investigators are also expecting a greater improvement in all those domains when participants are doing both interventions.

Objective 2: To evaluate the implementation strategy involving the virtual delivery of cognitive health interventions combined with a digital learning platform (E-Cog) to train mental health practitioners across multiple care settings. The investigators will assess how this strategy promotes the uptake of these cognitive health interventions across different mental health care settings. More specifically, the investigators will assess:

i) whether the E-Cog digital learning platform represents an effective educational strategy for implementation, ii) the contextual factors influencing the implementation of the two virtual interventions (i.e., potential barriers and facilitators to adoption) across sites, and iii) sustainability, the extent to which these interventions will be maintained within a service setting's ongoing operations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of affective or non-affective psychosis or related disorder;
* Follow-up and treatment by a clinician at one of the services mentioned above;
* Participants symptomatically stable and capable of using the online platforms and participating in intervention groups, as judged by their primary clinicians (i.e., psychiatrist, case manager);
* Participants must have access to a private space (i.e., a room where the participant can be alone) to ensure confidentiality for the group;
* Participants must be able to nominate an emergency contact and to agree to allow researchers to contact their clinician and/or emergency services in the event of an emergency during study procedures.

Exclusion Criteria:

* Intellectual disability;
* Hospitalization at the time of recruitment;
* Inability to speak or read English or French;
* High suicide risk as per evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Brief version of the Cambridge Neuropsychological Testing Automated Battery (CANTAB) score at the end of the intervention | Baseline to post (10 weeks)
  This brief version of the computerized battery assessing neurocognition provides z-scores (with zero indicating the mean of a group of values) for each MATRICS cognitive subdomain.
Change from Baseline Wechsler Memory Scale - Logical Memory (LM) subscale score at the end of the intervention | Baseline to post (10 weeks)
  In the LM I (maximum score=50), the two narrative stories (story A and story B) are verbally given and the examinee is required to immediately recall the stories as much as he/she can. In the LM II (maximum score=50), free recall of two stories is elicited after a 20 to 30-minute delay. Each correct detail was awarded with one score point. The 30 recognition questions (either yes or no) about the two stories are given subsequently to assess the recognition ability (maximum score=30).
Change from Baseline Brief Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS-B) score at the end of the intervention | Baseline to post (10 weeks)
  The SSTICS-B is a 14-item measure focusing on difficulties associated with core cognitive domains including memory, attention, executive functions and praxia. Each item is rated on a five-point Likert scale ranging from "never" to "very often" with higher scores suggesting more cognitive problems.
Change from Baseline Cognitive Motivation Scale (CMS) score at the end of the intervention | Baseline to post (10 weeks)
  Multidimensional scale for cognitive motivation assessing approach and withdrawal from cognitively challenging activities.
Change from Baseline Davos Assessment of Cognitive Biases Scale (DACOBS) score at the end of the intervention | Baseline to post (10 weeks)
  This questionnaire assesses cognitive biases through 42 items rated on a Likert scale from 1 (strongly disagree) to 7 (strongly agree).
Change from Baseline Beads task score at the end of the intervention | Baseline to post (10 weeks)
  In the beads task, participants see two jars full of beads of two colors. The beads in the jar have equal, but opposite ratios. One jar is chosen at random and kept secret from participants. As beads are drawn one at a time from the "secret" jar, participants must decide from which jar the beads are being drawn, or request to see more beads before deciding.
  In this task, the number of beads drawn before the participant makes a decision determines their tendency of "jumping to conclusion". Deciding with minimal "evidence" (less beads, or after the first bead is drawn) would indicate a higher tendency to jump to conclusions.
Change from Baseline bias against disconfirmatory evidence (BADE) image task score at the end of the intervention | Baseline to post (10 weeks)
  In this task, participants see partial line drawings of common objects, food or animals and are asked to whether they believe the full drawing corresponds to a word displayed below the image. The presence of a BADE bias in this task is represented by failing to modify an initial, erroneous hypothesis, once disconfirmatory evidence is provided.

SECONDARY OUTCOMES:
Change from Baseline Short version of the Positive And Negative Syndrome Scale (PANSS-6) score at the end of the intervention | Baseline to post (10 weeks)
  Through a semi-structured interview, the positive and negative symptomatology of schizophrenia is explored. In this reduced scale, the following symptoms are assessed: delusions, conceptual disorganization, hallucinations, flattened affect, passive social withdrawal, and poverty of speech.
Change from Baseline Brief Negative Symptom Scale (BNSS) score at the end of the intervention | Baseline to post (10 weeks)
  The Brief Negative Symptom Scale (BNSS) is a 13-item instrument measuring blunted affect, alogia, asociality, anhedonia, and avolition. All the items in the BNSS are rated on a 7-point (0-6) scale, with anchor points generally ranging from the symptom's being absent (0) to severe (6).
Change from Baseline Psychotic Symptom Rating Scales (PSYRATS) score at the end of the intervention | Baseline to post (10 weeks)
  The PSYRATS is comprised of 17 items inquiring about the specific dimensions of hallucinations and delusions, with each item being rated from 0 (absent) to 4 (severe).
Change from Baseline Emotional, and Social Loneliness Scale (OES) score at the end of the intervention | Baseline to post (10 weeks)
  It is a self-scale assessing the 3-item emotional loneliness and the 3-item social loneliness, two dimensions of the overarching loneliness concept.
Change from Baseline Self-Esteem Rating Scale - Short Form (SERS-SF) score at the end of the intervention | Baseline to post (10 weeks)
  The SERS consists of 20 items rated on a 7-point Likert scale, 10 scored positively and 10 negatively.
Change from Baseline Warwick-Edinburgh Mental Well-being Scale (WEMWBS) score at the end of the intervention | Baseline to post (10 weeks)
  The scale consists of 14 items covering both hedonic and eudaimonic aspects of mental health including positive affect (feelings of optimism, cheerfulness, relaxation), satisfying interpersonal relationships and positive functioning (energy, clear thinking, self acceptance, personal development, competence and autonomy).
Change from Baseline Questionnaire about the Process of Recovery (QRP) score at the end of the intervention | Baseline to post (10 weeks)
  The QPR is a 22 item self- report measure measuring the process of recovery from a psychotic disorder. The items are rated on a five-point Likert scale ranging from "strongly disagree" to "strongly agree".
Change from Baseline Personal and Social Performance scale (PSP) score at the end of the intervention | Baseline to post (10 weeks)
  The PSP scale assesses functioning across four dimensions (socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviours) with a maximum score of 100.

OTHER OUTCOMES:
Change from Baseline Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF) score at the end of the intervention | Baseline to post (10 weeks)
  this scale aims to assess satisfaction and frustration of the three basic psychological needs: competence, affiliation and autonomy. The items are reported on a scale ranging from 1 (completely disagree) to 7 (completely agree).
Change from Baseline Autonomous-Controlled Motivation for Intervention Questionnaire (ACMIQ) score at the end of the intervention | Baseline to post (10 weeks)
  Self-scale assessing motivational factors related to controlled and autonomous motivation.
Change from Baseline Health Care Climate Questionnaire (HCCQ) score at the end of the intervention | Baseline to post (10 weeks)
  The 6-item scale assesses motivational factors related to the therapists' perceived attributes (perceived support).
Change from Baseline MUSIC Cognitive Training Questionnaire score at the end of the intervention | Baseline to post (10 weeks)
  The MUSIC® Model of Motivation Inventory, Cognitive Training version (MMI-CT) is an 18-item self-report questionnaire that assesses motivation toward cognitive training. The questionnaire is divided into five scales namely empowerment, usefulness, success, interest and caring. Responses range from 1 (Strongly disagree) to 6 (Strongly Agree).
Program Sustainability Assessment Tool (PSAT) | Baseline to post (10 weeks)
  A 40-question assessment evaluating the sustainability capacity of a program by exploring 8 sustainability domains.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lepage, Principal Investigator — Douglas Mental Health University Institute
Locations (5):
- Canada (5):
  - Faculty of Medicine, University of British Columbia, Vancouver, British Columbia
  - Kingston Health Sciences Centre, Queen's University, Kingston, Ontario
  - Institute of Mental Health Research, University of Ottawa, Ottawa, Ontario
  - Ontario Shoares Centre for Mental Health Sciences, University of Toronto, Toronto, Ontario
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowie CR, Grossman M, Gupta M, Holshausen K, Best MW. Action-based cognitive remediation for individuals with serious mental illnesses: Effects of real-world simulations and goal setting on functional and vocational outcomes. Psychiatr Rehabil J. 2017 Mar;40(1):53-60. doi: 10.1037/prj0000189. Epub 2016 Apr 21. PMID 27100095
- [Background] Moritz S, Woodward TS. Metacognitive training in schizophrenia: from basic research to knowledge translation and intervention. Curr Opin Psychiatry. 2007 Nov;20(6):619-25. doi: 10.1097/YCO.0b013e3282f0b8ed. PMID 17921766
- [Background] Mendelson D, Thibaudeau E, Sauve G, Lavigne KM, Bowie CR, Menon M, Woodward TS, Lepage M, Raucher-Chene D. Remote group therapies for cognitive health in schizophrenia-spectrum disorders: Feasible, acceptable, engaging. Schizophr Res Cogn. 2021 Dec 6;28:100230. doi: 10.1016/j.scog.2021.100230. eCollection 2022 Jun. PMID 35242604
- [Derived] Au-Yeung C, Thai H, Best M, Bowie CR, Guimond S, Lavigne KM, Menon M, Moritz S, Piat M, Sauve G, Sousa AE, Thibaudeau E, Woodward TS, Lepage M, Raucher-Chene D. iCogCA to Promote Cognitive Health Through Digital Group Interventions for Individuals Living With a Schizophrenia Spectrum Disorder: Protocol for a Nonrandomized Concurrent Controlled Trial. JMIR Res Protoc. 2025 Apr 15;14:e63269. doi: 10.2196/63269. PMID 40233365